CLINICAL TRIAL: NCT00711867
Title: Intraoperative Warming: Comparison of Performance of the Dynatherm Medical vitalHeat™ Temperature Management System (vH2) and the Arizant Bair Hugger System
Brief Title: Comparison of Intraoperative Warming Devices
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Dynatherm Medical Inc. (Industry)
Responsible Party: Kent Weinmeister M.D., Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 07-003313
Record Dates: First submitted 2008-07-07; First posted 2008-07-09 (Estimated); Results first posted 2009-12-02 (Estimated); Last update posted 2009-12-15 (Estimated); Status verified 2009-12

CONDITIONS: Total Knee Arthroplasty

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- VH2 (Experimental): Dynatherm vitalHeat2 (VH2) temperature management system.
  Interventions: Device: VH2
- Bair Hugger (Active Comparator): Arizant Bair Hugger temperature management system.
  Interventions: Device: Bair Hugger

INTERVENTIONS:
Device: VH2 — Dynatherm vitalHeat2 (VH2) temperature management system.
  Arms: VH2
Device: Bair Hugger — Arizant Bair Hugger temperature management system.
  Arms: Bair Hugger

SUMMARY:
The sublingual (under the tongue) core temperature within 10 minutes of arrival in the post anesthesia care unit (PACU) for patients warmed with the Dynatherm vitalHeat2 (VH2) System under general anesthesia for total knee arthroplasty will be equivalent to that of patients warmed with the Arizant Bair Hugger System.

ELIGIBILITY:
Inclusion Criteria:

* Initial total knee arthroplasty.
* Expected duration of surgery at least 2 hours.
* General anesthesia.
* American Society of Anesthesiologists (ASA) classification I-III.
* Age >= 18 years.

Exclusion Criteria:

* Skin abrasion at the device application site.
* History of peripheral vascular disease.
* History of allergic skin conditions of the upper extremities.
* History of malignant hyperthermia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2008-07; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kent Weinmeister, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Phoenix, Arizona, United States

REFERENCES:
- [Derived] Trentman TL, Weinmeister KP, Hentz JG, Laney MB, Simula DV. Randomized non-inferiority trial of the vitalHEAT temperature management system vs the Bair Hugger warmer during total knee arthroplasty. Can J Anaesth. 2009 Dec;56(12):914-20. doi: 10.1007/s12630-009-9199-2. Epub 2009 Sep 25. PMID 19779953

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited sequentially and assigned to vitalHeat2 (VH2) or Bair Hugger temperature management at random in a 1:1 ratio.
Pre-assignment Details: 75 consented. 9 cancelled surgery or were rescheduled. 36 assigned to VH2 and 30 assigned to Bair Hugger. 6 excluded from VH2 group after randomization (2 vacuum not established, 2 research staff not available, 2 arterial line used). 5 excluded from Bair Hugger group after randomization (4 laryngeal mask airway used, 1 epidural anesthesia used).
Groups:
- VH2 Temperature Management: Dynatherm vitalHeat2 (VH2) temperature management system.
- Bair Hugger Temperature Management: Arizant Bair Hugger temperature management system.
Period: Overall Study
Arm/Group | VH2 Temperature Management | Bair Hugger Temperature Management
Started | 30 | 25
Completed | 25 (2 received additional warming. 3 missing primary measure.) | 21 (3 received additional warming. 1 missing primary measure.)
Not Completed | 5 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | VH2 Temperature Management | Bair Hugger Temperature Management | Total
Number analyzed (Participants) | 30 | 25 | 55
Age Continuous [Mean (Standard Deviation); unit: years] | 68.9 (11.4) | 67.0 (9.4) | 68.0 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 13 | 31
  Male | 12 | 12 | 24

OUTCOME MEASURES:

1. Primary Outcome: Sublingual Temperature.
Time Frame: Within 10 minutes of arrival in PACU
Population: Per protocol.
Measure: Mean (Standard Deviation); unit: C
Arm/Group | VH2 Temperature Management | Bair Hugger Temperature Management
Number analyzed (Participants) | 25 | 21
C | 36.38 (0.38) | 36.73 (0.29)
Statistical Analysis 1: Comparison: VH2 Temperature Management vs Bair Hugger Temperature Management; H0: Mu_VH - Mu_BH <= -0.5 C; Test type: Non-Inferiority or Equivalence — The non-inferiority margin was defined as -0.5 C; t-test, 2 sided; Mean Difference (Final Values) = -0.34, 95% CI [-0.55 to -0.14]

ADVERSE EVENTS:
Arm/Group | VH2 Temperature Management | Bair Hugger Temperature Management
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/25
Other Adverse Events (participants affected / at risk) | 0/30 | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less